CLINICAL TRIAL: NCT06397287
Title: Standardized Collection of Patient Reported Outcomes (PROs) in Everyday Clinical Practice
Brief Title: PROM Project Urology
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-405 ex 22/23
Record Dates: First submitted 2024-03-28; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Surgery; Urologic Diseases; Urologic Cancer
MeSH Terms: conditions — Urologic Diseases; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of patients undergoing sugery — All patients undergoing urological surgery or treatment receive standardized questionnaires on quality of life, satisfaction, pain and physical recovery. Indication-specific, individual pathways are set up,

SUMMARY:
All patients undergoing urological surgery or treatment should receive standardized questionnaires on quality of life, satisfaction, pain and physical recovery. Indication-specific, individual pathways are set up, for example, for patients with localized prostate cancer, benign prostate enlargement, bladder dysfunction or erectile dysfunction. In combination with the clinical data, the PROM data should help to improve the quality of the results and, if necessary, adapt treatment pathways to patient needs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated at the Department of Urology
2. ≥18 years of age
3. Active Mail-account, use of smartphone/tablet/PC
4. Written informed consent

Exclusion Criteria:

- Patients who cannot give written consent and/or do not have digital competence (e.g. no active e-mail account)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Specific urologic diseases are dependent on gender
Study Population: Patients treated at the Department of Urology
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2045-09-05 (Estimated); Study Completion 2045-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in functional treatment outcome in patients with prostate cancer, assessed by EPIC-26: (Expanded Prostate cancer Index Composite) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment EPIC-26 score: max 100 points; greater values indicate improved functional outcomes
Change in health-related quality of life (PROMIS-10: Patient-Reported Outcomes Measurement Information System) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. PROMIS-10 max 50 points; greater values indicate healthier status
Change in pain: Brief Pain Inventory (BPI) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. BPI: max. 11 points; greater values indicate worse outcome
Change in erectile function (IIEF: International Index of Erectile Function) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. IEF: 0-25 points; greater values indicate better ercetile function
Change in bladder function/micturition (IPSS: International Prostate Symptom Score) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. IPSS: score 0-35; greater values indicates increased symptom severity
Change in bladder function/micturition (OAB-SF: Overactive Bladder Questionnaire, short form) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. OAB-SF: score 0 - 16; score with greater values indicates increased symptom severity
Change in bladder function/micturition (ICIQ-UI: International Consultation on Incontinence Questionnaire-Urinary Incontinence) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. ICIQ-UI: score 0-21; greater values indicate worse urinary incontinence
Change in pelvic pain (NHS-CPSI: Chronic prostatits symptom index) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Electronically recorded Patient Reported Outcomes (PROs) are captured for each patient depending on the condition and surgery/treatment. NHS-CSI: 0-43 points; greater values indicate worse outcomes

SECONDARY OUTCOMES:
patient characteristics: age | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Clinical parameters are captured for each patient undergoing sugery
patient characteristics:comorbidities | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Clinical parameters are captured for each patient undergoing sugery
patient characteristics: medication (name, type, dose, interval) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Clinical parameters are captured for each patient undergoing sugery
patient characteristics: disease-specific data (tumor histology, oncologic status) | Data collection/follow-up: day - 1 before surgery, 2 to 10 days host surgery, after 3, 6, 12 months, annually 2 to 10 years
  Clinical parameters are captured for each patient undergoing sugery
Perioperative data: duration of sugery (minutes) | during surgery, surgery time depending on the disease (30 minutes to 4 hours)
  Perioperative data are captured for each patient undergoing sugery
Perioperative data: blood loss (ml) | during surgery, surgery time depending on the disease (30 minutes to 4 hours)
  Perioperative data are captured for each patient undergoing sugery
Perioperative data: transfusion (ml | during surgery, surgery time depending on the disease (30 minutes to 4 hours)
  Perioperative data are captured for each patient undergoing sugery
Perioperative data: length of hospital stay (days) | depending on the disease and following surgery (1 to 10 days)
  Perioperative data are captured for each patient undergoing sugery

CONTACTS AND LOCATIONS:
Locations (1):
- Röthl Martina Anna, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided